CLINICAL TRIAL: NCT01519297
Title: Preeclampsia: A Marker for Future Cardiovascular Risk in Women
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Pending funding
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ellen W. Seely, M.D., Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PP PE 2012
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Preeclampsia; Pregnancy Induced Hypertension
Keywords: Preeclampsia; Pregnancy Induced Hypertension
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced | interventions — Irbesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm intervention (Other): Irbesartan 150 mg orally for one dose
  Interventions: Drug: Irbesartan

INTERVENTIONS:
Drug: Irbesartan — 150mg orally for one dose

SUMMARY:
This study will compare blood vessel and hormone differences between women who have a history of a pregnancy complicated by preeclampsia or high blood pressure, and women who have a history of uncomplicated pregnancy in the last 10 years. The investigators hypothesize that postpartum women with history of preeclampsia will have altered blood vessel function and abnormal hormone levels compared with postpartum women with history of uncomplicated pregnancy.

This study will take place over the course of 2 weeks. Each subject will be assessed on a fixed low-salt diet and a fixed high-salt diet. Subjects will have 2 non-invasive blood vessel imaging tests and fasting blood draws.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female premenopausal volunteers, with regular menstrual cycles (at least 8 cycles per year)
2. Age 21 to 50 years
3. Systolic blood pressure <140 and >90 mmHg and diastolic blood pressure <90 and >60 mmHg at the screening visit
4. Body mass index < 35 kg/m2
5. History of normotensive pregnancy or history of preeclamptic or hypertensive pregnancy within the last 10 years
6. No clinically significant abnormalities on screening tests (complete blood count, serum electrolytes, liver enzymes, thyroid stimulating hormone, urinalysis, and electrocardiogram)

Exclusion Criteria:

1. Current pregnancy
2. Lactation
3. Elevated blood pressure (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg)
4. Current diagnosis of hypertension
5. Current diagnosis of diabetes mellitus
6. Personal history of coronary disease, stroke and kidney disease
7. Use of prescription medications (with the exception of stable thyroid hormone replacement dose) within 2 weeks of study
8. Use of oral contraceptives or other hormone therapy within 3 months of study;
9. Renal impairment (estimated GFR<60)
10. Active liver disease (AST, ALT, alkaline phosphatase > 1.5 times normal);
11. Current smoking, defined as smoking within the 6 months before the screening visit
12. Current or past recreational drug use

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Vascular function | 60 minutes
  Assess vascular function after administration of an angiotensin receptor blocker.

SECONDARY OUTCOMES:
Hormonal measurements | 60 minutes
  Assess hormone levels pertaining to the renin-angiotensin system after administration of irbesartan.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen W Seely, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States